CLINICAL TRIAL: NCT04558905
Title: Impact of a Hybrid Medical Care Model (Face-to-face Medical Visits Alternating With Video Medical Consultations) in the Rheumatoid Arthritis Patient-reported-outcomes Measures: A Non-inferiority Study
Brief Title: Impact of a Hybrid Medical Care Model in the Rheumatoid Arthritis Patient-reported-outcomes Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Medical Sciences and Nutrition, Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Virginia Pascual Ramos, Rheumatologist, National Institute of Medical Sciences and Nutrition, Salvador Zubiran
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: IRE-3438 20221
Record Dates: First submitted 2020-09-10; First posted 2020-09-22 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Rheumatoid Arthritis; Telehealth
Keywords: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: This a non-inferiority and cross-over study, with a planned follow-up of 16 months, with 2 intervention arms:
  Intervention 1: Patients assigned to 6 months of usual medical care model, followed by 4 months of a control period, and finally 6 months of hybrid medical care model.
  Intervention 2: Patients assigned to 6 months of hybrid medical care model, followed by 4 months of a control period, and finally 6 months of usual medical care model.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Medical Care Model (Active Comparator): All the patients will receive face-to-face medical visits
  Interventions: Other: Face-to-face medical visits
- Hybrid Medical Care Model (Experimental): The patients will receive alternating face-to-face medical visits and video medical consultations
  Interventions: Other: Alternating face-to-face medical visits and video medical consultations

INTERVENTIONS:
Other: Face-to-face medical visits — Face-to-face medical visits
  Arms: Usual Medical Care Model
Other: Alternating face-to-face medical visits and video medical consultations — Alternating face-to-face medical visits and video medical consultations
  Arms: Hybrid Medical Care Model

SUMMARY:
The COVID-19 outbreak has affected health care of patients with rheumatic diseases; telemedicine might help to assist patients.

The primary objective is to determine if a hybrid medical care model, which consists of alternating face-to-face medical visits and video medical consultations, is not inferior, in terms of the Patient Reported Outcomes measures (PROMs), to the face-to-face medical care model, among rheumatoid arthritis (RA) outpatients. We also aim to investigate if adherence to RA-related treatment (considered a surrogate of patient´s education) might be improved when patients are re-integrated to the health care system, irrespective of the health care model.

In Mexico, COVID-19 pandemic still uncontrolled. Our Institution provides health care to 1500 RA patients/year and up to August 2020, it is estimated that 500 RA patients might be affected, which is our target audience. Reinstalling institutional health care provision is challenging.

This a non-inferiority, cross-over study, with 2 intervention arms. Patients will be randomized to 1. Six months of usual medical care model, followed by 4 months of a control period, and 6 months of hybrid medical care model, or 2. Six months of hybrid medical care model, followed by 4 months of a control period, and 6 months of usual medical care model.

The following PROMs will be assessed at specific time points: disease activity/disease severity (RAPID-3), disability (HAQ-DI), quality of life (WHOQOL-BREF), patient satisfaction with the medical care model (questionnaire locally developed), patient´s adherence to medical care (missed scheduled visits) and patient´s adherence to RA-related treatment (the Compliance-Questionnaire).

DETAILED DESCRIPTION:
This a non-inferiority and cross-over study, with a planned follow-up of 16 months, with 2 intervention arms:

Intervention 1: Patients assigned to 6 months of usual medical care model, followed by 4 months control period, and finally 6 months of hybrid medical care model.

Intervention 2: Patients assigned to 6 months of hybrid medical care model, followed by 4 months control period and finally 6 months of usual medical care model.

Specific objectives are as follows:

Primary objectives

1. To compare the mean disease activity of RA patients (as measured per RAPID-3), after 6 months since study entry, between patients assigned to intervention 1 and patients assigned to intervention 2.
2. To compare the RA patient´s quality of life (as measured per WHOQOL-BREF) and RA patient's disability (as measured per HAQ-DI) after 6 months since study entry, between patients assigned to intervention 1 and patients assigned to intervention 2.

Secondary objectives:

1. At the end of the complete follow-up period, for each patient, to compare the cumulative RA disease activity during the 6 months period where patients received usual medical care model, with the cumulative disease activity during the 6 months period where patients received hybrid medical care model.
2. At the end of the complete follow-up period, for each patient, to compare patient´s satisfaction with usual medical care model and patient´s satisfaction to hybrid medical care model.
3. At the end of the complete follow-up period, for each patient, to compare patient´s adherence to the usual medical care model with patient´s adherence to hybrid medical care model.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA diagnosis according to their primary rheumatologist
* With at least six months of follow-up (up to March 2020) at the outpatient clinic
* Who agree to participate

Exclusion Criteria:

* Patients lost to follow-up from the outpatient clinic before March 2020
* Patients with no access to a mobile device during their study participation
* Patients with severe cognitive, visual and hearing impairment
* Patients on palliative care because of comorbid condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Rheumatoid arthritis patient´s disease activity | During the 16 months of follow up, the evaluations will be in each medical visits (in both medical care models)
  The disease activity measured by a RAPID-3 instrument
Rheumatoid arthritis patient´s quality of life | During the 16 months of follow up, the evaluations will be in each medical visits (in both medical care models)
  Quality of life measured by a WHOQOL-BREF instrument
Rheumatoid arthritis patient's disability | During the 16 months of follow up, the evaluations will be in each medical visits (in both medical care models)
  Disability measured by a HAQ-DI instrument

SECONDARY OUTCOMES:
Satisfaction with medical care | During the 16 months of follow up, the evaluations will be in each medical visits (in both medical care models)
  Questionnaire locally developed
Patient´s adherence to medical care | During the 16 months of follow up, the evaluations will be in each medical visits (in both medical care models)
  Number of missed scheduled visits

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pascual-Ramos, Dr., Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: No